CLINICAL TRIAL: NCT00342888
Title: A Case-Control Study of Pesticides and Childhood Leukemia
Brief Title: Case-Control Study of Pesticides and Childhood Leukemia
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902030; 02-C-N030; NCT00556985 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-10

CONDITIONS: Leukemia
Keywords: Childhood Cancer; Pesticides; Polychlorinated Biphenyls; Organochlorines; Polybrominated Diphenyl Ethers; Natural History
MeSH Terms: conditions — Leukemia; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Childhood Leukemia Cases: Cases were diagnosed at 9 hospitals in Northern California
- Matched Controls: Controls were matched on age, gender and race/ethnicity from birth certificates in Northern California

SUMMARY:
Childhood leukemia is the most common type of childhood cancer and its etiology is largely unknown. Most case-control studies of childhood leukemia have reported elevated risks among children whose parents were occupationally exposed to pesticides or who used pesticides in the home or garden. Investigators at the University of California at Berkeley (UCB) conducted a case-control study of childhood leukemia in 35 counties in the San Francisco Bay area and the agricultural Central Valley of California. A major focus of the UCB study is to evaluate whether household or occupational exposure to pesticides increases the risk of childhood leukemia. Our collaboration provided additional funding to collect carpet dust samples for the measurement of pesticides and other chemicals. For 470 participants, we attempted to collect carpet dust using a special high volume small surface sampler (HVS3) vacuum and by taking dust from participants vacuum cleaner. As of July 2006, dust samples will be collected only from participant's vacuum cleaner. Samples were collected at a home visit approximately 3-6 months after the first in-person interview. We will also provide support for mapping of the crops (i.e., determining crop field boundaries and crop species) within 1200 meters (3/4 mile) of residences so that the residential proximity to agricultural fields treated with pesticides can be determined. We will conduct the epidemiologic analysis of pesticide and other chemical levels in carpet dust and risk of childhood leukemia. We will also evaluate whether residential proximity to agricultural pesticide use is associated with risk of leukemia. Further, we will conduct an Exposure Pilot Study that will include a subset of the study population. Two components of the Pilot Study will evaluate how well a used vacuum bag and a window sill wipe predict pesticide and other chemical concentrations in carpet dust samples collected with the more complicated HVS3 vacuum method. The third component will compare pesticides detected in carpet dust with pesticides predicted by geographic proximity to agriculture.

DETAILED DESCRIPTION:
Childhood leukemia is the most common type of childhood cancer and its etiology is largely unknown. Most case-control studies of childhood leukemia have reported elevated risks among children whose parents were occupationally exposed to pesticides or who used pesticides in the home or garden. Investigators at the University of California at Berkeley (UCB) conducted a case-control study of childhood leukemia in 35 counties in the San Francisco Bay area and the agricultural Central Valley of California. A major focus of the UCB study was to evaluate whether household or occupational exposure to pesticides increases the risk of childhood leukemia. Our collaboration provided additional funding to collect carpet dust samples for the measurement of pesticides and other chemicals. For 470 participants, we attempted to collect carpet dust using a special high volume small surface sampler (HVS3) vacuum and by taking dust from participants vacuum cleaner. As of July 2006, dust samples were collected only from participant's vacuum cleaner. Samples were collected at a home visit approximately 3-6 months after the first in-person interview. We also provided support for mapping of the crops (i.e., determining crop field boundaries and crop species) within 1200 meters (3/4 mile) of residences so that the residential proximity to agricultural fields treated with pesticides can be determined. We will conduct the epidemiologic analysis of pesticide and other chemical levels in carpet dust and risk of childhood leukemia. We will also evaluate whether residential proximity to agricultural pesticide use is associated with risk of leukemia. Further, we will conduct an Exposure Pilot Study that will include a subset of the study population. Two components of the Pilot Study will evaluate how well a used vacuum bag and a window sill wipe predict pesticide and other chemical concentrations in carpet dust samples collected with the more complicated HVS3 vacuum method. The third component will compare pesticides detected in carpet dust with pesticides predicted by geographic proximity to agriculture.

ELIGIBILITY:
* INCLUSION CRITERIA:

All cases and controls were selected from participants in the UCB case-control study who have completed the Tier I interview.

Study population is limited to children.

All races and ethnicities will be included in the study.

Tier I:

The cases eligible for participation in Tier I of the UCB study of all newly diagnosed cases of childhood leukemia 0-14 years old resident in 35 counties in San Francisco Bay Area and the Central Valley

Further inclusion criteria are no prior cancer diagnosis and at least one English or Spanish speaking parent.

Tier II:

Tier II participants will be selected from cases and controls that complete the Tier I interview. Cases (and their match controls), aged 0-7, diagnosed from December 1, 1999 through 2003, and who still reside at the home where they were living ate the diagnosis date, will be eligible for the Tier II interview.

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Population-based study of childhood leukemia in 35 counties in northern and central California. Cases were diagnosed at 9 hospitals in these counties and controls were residents of California selected from California birth certificates and matched to cases by birth date, gender, race/ethnicity
Sampling Method: Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2001-10-30 (Actual)

PRIMARY OUTCOMES:
odds ratios for exposures to environmental contaminants and other factors related to childhood leukemia. | Data analysis still ongoing
  childhood leukemia
factors associated with concentrations of chemicals including pesticides and persistent organochlorines in house dust samples | Data analysis still ongoing
  concentrations of the chemicals

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Jones, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Background] Metayer C, Colt JS, Buffler PA, Reed HD, Selvin S, Crouse V, Ward MH. Exposure to herbicides in house dust and risk of childhood acute lymphoblastic leukemia. J Expo Sci Environ Epidemiol. 2013 Jul;23(4):363-70. doi: 10.1038/jes.2012.115. Epub 2013 Jan 16. PMID 23321862
- [Background] Deziel NC, Rull RP, Colt JS, Reynolds P, Whitehead TP, Gunier RB, Month SR, Taggart DR, Buffler P, Ward MH, Metayer C. Polycyclic aromatic hydrocarbons in residential dust and risk of childhood acute lymphoblastic leukemia. Environ Res. 2014 Aug;133:388-95. doi: 10.1016/j.envres.2014.04.033. Epub 2014 Jun 17. PMID 24948546
- [Background] Ward MH, Colt JS, Metayer C, Gunier RB, Lubin J, Crouse V, Nishioka MG, Reynolds P, Buffler PA. Residential exposure to polychlorinated biphenyls and organochlorine pesticides and risk of childhood leukemia. Environ Health Perspect. 2009 Jun;117(6):1007-13. doi: 10.1289/ehp.0900583. Epub 2009 Jan 27. PMID 19590698